CLINICAL TRIAL: NCT06343246
Title: The Effect of Functional Inspiratory Muscle Training on Exercise Capacity, Peripheral Muscle Strength in Patients With Hypertension
Brief Title: Functional Inspiratory Muscle Training in Patients Diagnosed With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Irem Hüzmeli, Assistant Prof. PhD, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MustafaKemalU
Record Dates: First submitted 2024-03-19; First posted 2024-04-02 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Hypertension,Essential
Keywords: exercise; peripheric muscle strenght; inspiratory muscle training; high blood pressure; functionality
MeSH Terms: conditions — Essential Hypertension; Motor Activity; Hypertension

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Functional IMT Group (Experimental): Functional IMT Group (n:15) : will recieve functional inspiratory muscle training (exercise + 50% of MIP)
  Interventions: Device: Inspiratory muscle training with device
- IMT Group (Active Comparator): IMT Group I (n:15): will recieve inspiratory muscle training (50% of MIP )
  Interventions: Device: Inspiratory muscle training with device
- Control group (Experimental): Control group (n:15): will recieve breathing exercises training
  Interventions: Device: Inspiratory muscle training with device

INTERVENTIONS:
Device: Inspiratory muscle training with device — : A randomized, controlled three-arm study. Forty-five patients with HT randomized three group: Group 1 will receive IMT (7 days/8 weeks) with function and POWERbreathe® Classic LR device, group 2 will reviece only IMT with 50 % maximal inspiratory pressure (MIP), n: 15) and control group will recieve breathing exercises(7 days/8 weeks).

SUMMARY:
This study was planned to investigate the effectiveness of combined exercise training, that is, functional inspiratory muscle training, with breathing exercises to be applied with a portable, easy-to-use respiratory muscle strengthening device, on exercise capacity and peripheral muscle strength.

DETAILED DESCRIPTION:
Forty-five Individuals will be randomly divided into three groups:

Functional IMT Group (n:15): will receive functional inspiratory muscle training (exercise + 50% of MIP) IMT Group I (n:15): will recieve inspiratory muscle training (50% of MIP ) Control group (n:15): will recieve breathing exercises training

ELIGIBILITY:
Inclusion Criteria:

1. Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg,
2. It will include both male and female subjects aged ≥18 and <80 years with a previous diagnosis of essential hypertension.
3. Subjects receiving no pharmacological treatment or receiving only thiazide diuretics
4. Those with a body mass index <30 kg/m2 Those who engage in <150 minutes of moderate or intense physical activity per week, according to the 5th International Physical Activity Survey

Exclusion Criteria:

1. Blood pressure ≥160 / 100 mmHg
2. Severe dyspnea; diabetes; orthopedic, musculoskeletal, or fitness limitations;
3. Major physiological crises;
4. A current or past history of deep venous thrombosis; History of myocardial infarction or stroke within the 5th year or 6 months ago;

6. Congestive heart therapy; 7. Unstable angina; 8. or lung disease of any etiology (including asthma and chronic obstructive pulmonary disease); 9. Active smokers 10. Patients under 18 years of age 11. Pregnant women 12. Those with Active Infection 13. Those with Known Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change of the exercise capacity from baseline to 8 week | from baseline to 8 week
  Exercise capacity was evaluated with the 6-Minute Walk Test (6MWT). ATS (American Thoracic Society) criteria were taken into consideration and the subjects rested for at least half an hour before starting the test. Participants walked briskly at their own walking pace for 6 minutes on a 30-meter straight corridor. The distance reached at the end of the test was recorded in meters.
Change of the peripheral muscle strenght from baseline to 8 week | from baseline to 8 week
  Peripheral muscle strength and hand grip strength were evaluated with a portable dynamometer and the values obtained were recorded in Newton (N)/kgF/Pascal. Peripheral muscle strength was measured seated, employing a hand-held dynamometer (JTECH Power Track Commander, Baltimore, MD, USA). This device, known for its portability and cost-effectiveness, serves as an alternative to isokinetic machines and offers greater sensitivity in detecting changes in muscle strength compared to manual muscle tests.
  Respiratory muscle strength 'maximum inspiratory pressure (MIP) and expiratory pressure (MEP)' will calculate with a portable, electronic mouth pressure measuring device.
change of the upper extremity exercise capacity from baseline to 8 week | from baseline to 8 week
  6PBRT is a test used to evaluate unsupported upper extremity exercise capacity. Participants will be asked to sit in an adjustable-height chair. The pegboard will be placed within arm's reach of the person. Participants will be asked to attach a total of 20 rings, 32 rings, 10 on each iron rod, located at both shoulder levels, to the iron rods 20 centimeters above, as quickly as possible, using both arms simultaneously, for six minutes, and then to attach and remove them again to the iron rods below.

SECONDARY OUTCOMES:
change of the postural balance from baseline to 8 week | from baseline to 8 week
  Timed Up and Go test (TUG): It measures the time it takes for the patient to get up from the chair, walk 3 m, turn around and sit down in the same chair again. The TUG test is a simple test used to evaluate postural mobility
change of the physical activity from baseline to 8 week | from baseline to 8 week
  Physical activity level was measured with the International Physical Activity Questionnaire (IPAQ). In this questionnaire, which provides information about the time spent in sitting, walking, moderately vigorous activities, and vigorous activities, the criterion for evaluating all activities is that each activity is performed for at least 10 minutes at a time.
change of the quality of life from baseline to 8 week | from baseline to 8 week
  SF-36 survey. In this scale, where health is examined in eight components, higher scores indicate a better level of health. SF-36 scale; physical functionality (limitation in physical activity due to health problems), physical role limitation in daily living activities due to health problems), bodily pain, general health (evaluation of the person's general health), vitality , general mental health, social functionality and emotional role (limitation in daily living activities due to mental health problems). The SF-36 scale is scored out of 100 points, and the scores vary between 0 and 100 points for each component.
change of the Fev1/Fvc | from baseline to 8 week
  Pulmonary function test will measure with a portable spirometer (SPIROBANK II® Moggiolino, Rome-Italy). The best of 3 technically acceptable maneuvers with 95% agreement will select and record

CONTACTS AND LOCATIONS:
Overall Officials: İrem Hüzmeli, Principal Investigator — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Antakya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huzmeli I, Katayifci N, Abay B, Akkus O, Ozer AY. The effectiveness of functional inspiratory muscle training on exercise capacity and peripheral muscle strength in patients with essential hypertension: a three-arm randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 Feb 28;17(1):29. doi: 10.1186/s13102-025-01082-w. PMID 40022256